CLINICAL TRIAL: NCT03268447
Title: Lactobacillus Plantarum P8 for Its Brain Health Promotion Potential
Acronym: P8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Beijing Scitop Bio-Tech Shareholding Co.Ltd. (Unknown)
Responsible Party: Principal Investigator, Min-Tze LIONG, Professor Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USM/JEPeM/16050195
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Placebo and P8 will be administered via a parallel design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum P8 (Active Comparator): Intervention consists of daily administration of 2g probiotic Lactobacillus plantarum P8, administered daily at a fixed dosage of 10 log CFU/sachet/day and continue for 12 weeks.
  Interventions: Dietary Supplement: Lactobacillus plantarum P8
- Placebo (Placebo Comparator): Intervention consists of daily administration of 2g placebo (no probiotic bacteria), administered daily and continue for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum P8 — This project aims to study the benefits of probiotics namely Lactobacillus plantarum P8 for brain health benefits primarily to alleviate stress, among adults in Malaysia aged from 18-60 years.
  Other Names: P8
  Arms: Lactobacillus plantarum P8
Dietary Supplement: Placebo — This project aims to study the benefits of probiotics namely Lactobacillus plantarum P8 for brain health benefits primarily to alleviate stress, among adults in Malaysia aged from 18-60 years.
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Lactobacillus plantarum P8 for brain health properties, primarily alleviation of stress, among adults in Malaysia aged from 18 to 60 years.

DETAILED DESCRIPTION:
The emerging concept of gut-brain-axis has been implying that gut health plays a pivotal role in maintaining brain health4. Probiotics have entered the picture in promoting gut health for better brain health. Probiotic can be defined as "live microorganisms that grant health effects to the host if consumed in sufficient amounts". Lactobacilli, as one of the largest genera for probiotic microorganisms have been researched to alleviate stress, anxiety and/or depression disorders.

L. plantarum P8 was isolated from traditionally fermented sour milk samples collected from herdsmen in Wulatezhongqi grassland, Bayannaoer, Inner Mongolia, China. L. plantarum P8 was selected as it was the best among 347 other Lactobacillus strains with excellent tolerance to gastric acid, intestinal fluid and bile salt of the digestive system. P8 is incorporated and sold in the market of China, Taiwan and Singapore in a variety of products, ranging from dairy (yoghurt and fermented milk), health supplements to pet foods. P8 is patented in China and also awarded by the Chinese government as a functional probiotic. Two human clinical trials have shown that the administration of P8 at a concentration of 10 log CFU/day for 4-weeks, improved gastrointestinal health of adults subjects via increasing the population of beneficial gut microbiota accompanied by decreasing gut opportunistic pathogens, increasing fecal levels of secretory immunoglobulin-A and short chain fatty acids.

Thus, with evidence from other studies supporting the stress-alleviation effects of lactobacilli and the current gut modulation properties of P8, we believe that L. plantarum P8 could exert stress alleviation potentials as well.

P8 has confirmed its safety for consumption, and for this intervention, it will be produced under ISO9001 and HALAL in China. HALAL certification is provided by ARA HALAL Development Services Center Inc. (ARA), which is recognized by JAKIM, Malaysia, an organization that oversees the implementation of Halal requirement in Malaysia.

A total number of 176 healthy adults from age 18 -60 years old will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* 18-60 years old
* No severe illness
* BMI within a healthy range
* Score between 13 -20 (moderate stress level) on Cohen's Perceived Stress Scale (PSS)
* Willing to commit throughout the experiment

Exclusion Criteria:

* Type-1 diabetes (one of the main metabolite of Lactobacillus is acetic acid. Acetic acid has been reported to affect lipid metabolism in the liver and fat digestion in the pancreas in animal studies, and has been applied in obesity studies)
* Long term medication due to certain severe illness (certain medications may interfere with the survivability of Lactobacillus in the gut, for example the interactions between probiotics and warfarin
* HIV/AIDS (there has been no substantial data on the detrimental effects of probiotics on AIDS patients. However, AIDS patient may be immune-compromised in the sense of "leaky gut" that may lead to bacterial translocation, including translocation of Lactobacillus outside the gut environment, into the blood stream)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency (there has been no substantial data on the detrimental effects of probiotics on G6PD deficiency people. However, certain strains of probiotics have been reported to benefit RBC irregularity disorders such as spur cells formation. One of the main mechanisms, involve the alteration of RBC membrane. Although this is a benefit, we are unsure of the effects on G6PD deficiency people, with weaker RBC).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) Scores | 12 weeks
  Stress Questionnaires for the determination of stress (low, moderate, high)

SECONDARY OUTCOMES:
Fecal microbiota profiling | 12 weeks
  Deoxyribonucleic acid (DNA) sequencing of fecal samples to compare DNA sequences of the different microbiota between adult participants taking P8 vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Min Tze Liong, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- School of Industrial Technology, Universiti Sains Malaysia, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
General grouping data only

REFERENCES:
- [Background] Kwok LY, Guo Z, Zhang J, Wang L, Qiao J, Hou Q, Zheng Y, Zhang H. The impact of oral consumption of Lactobacillus plantarum P-8 on faecal bacteria revealed by pyrosequencing. Benef Microbes. 2015;6(4):405-13. doi: 10.3920/BM2014.0063. Epub 2015 Feb 12. PMID 25653153
- [Background] Wang L, Zhang J, Guo Z, Kwok L, Ma C, Zhang W, Lv Q, Huang W, Zhang H. Effect of oral consumption of probiotic Lactobacillus planatarum P-8 on fecal microbiota, SIgA, SCFAs, and TBAs of adults of different ages. Nutrition. 2014 Jul-Aug;30(7-8):776-83.e1. doi: 10.1016/j.nut.2013.11.018. Epub 2013 Dec 4. PMID 24984992
- [Derived] Lew LC, Hor YY, Yusoff NAA, Choi SB, Yusoff MSB, Roslan NS, Ahmad A, Mohammad JAM, Abdullah MFIL, Zakaria N, Wahid N, Sun Z, Kwok LY, Zhang H, Liong MT. Probiotic Lactobacillus plantarum P8 alleviated stress and anxiety while enhancing memory and cognition in stressed adults: A randomised, double-blind, placebo-controlled study. Clin Nutr. 2019 Oct;38(5):2053-2064. doi: 10.1016/j.clnu.2018.09.010. Epub 2018 Sep 19. PMID 30266270